CLINICAL TRIAL: NCT00767962
Title: A Prospective Randomised Study of Efficacy, Safety and Costs of Talc Pleurodesis Under Medical Thoracoscopy and Pleurodesis Under Video-assisted Thoracoscopy Surgery for Recurrent Primary Spontaneous Pneumothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-A00342-51
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Pneumothorax
Keywords: recurrent primary spontaneous pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): talc pleurodesis under medical thoracoscopy
  Interventions: Other: talc pleurodesis under medical thoracoscopy
- 2 (Other): pleurodesis under video-assisted thoracoscopy surgery
  Interventions: Other: pleurodesis under video-assisted thoracoscopy surgery

INTERVENTIONS:
Other: talc pleurodesis under medical thoracoscopy — talc pleurodesis under medical thoracoscopy for recurrent primary spontaneous pneumothorax
  Arms: 1
Other: pleurodesis under video-assisted thoracoscopy surgery — pleurodesis under video-assisted thoracoscopy surgery for recurrent primary spontaneous pneumothorax
  Arms: 2

SUMMARY:
Treatment of recurrent primary spontaneous pneumothorax remains controversial and many therapeutic options exist. The aim of this study is to compare pleural symphysis by talc poudrage during medical thoracoscopy and surgical management combining pleural abrasion and blebs or bullae resection for treatment of recurrent primary spontaneous pneumothorax.

DETAILED DESCRIPTION:
Treatment of recurrent primary spontaneous pneumothorax remains controversial and many therapeutic options exist. What is the best technical option : treatment of the lung and the parietal pleura or treatment of the pleura with pleural symphysis ? Talc pleurodesis performed during medical thoracoscopy and resection of blebs or bullae associated with pleural abrasion during surgical thoracoscopy (or video-assisted thoracic surgery) are the most usual methods. These two procedures have never been compared in a prospective trial. The aim of this study is to compare pleural symphysis by talc poudrage during medical thoracoscopy and surgical management combining pleural abrasion and blebs or bullae resection for treatment of recurrent primary spontaneous pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* Subjects :both sexes, who the age is included between 18 years and 55 years;
* Presenting a recurrence homolaterale or controlaterale of a primary spontaneous pneumothorax;
* Presenting a bilateral primary spontaneous pneumothorax
* Presenting a failure of a manual inhalation for a primary spontaneous pneumothorax;
* Presenting a persistent superior bullage at 48 am after a thoracic drainage for a spontaneous pneumothorax
* Presenting a persistent superior bullage at 48 am after a thoracic drainage for a primary spontaneous pneumothorax;
* Presenting a persistent superior unsticking at 48 am after a thoracic drainage for a primary spontaneous pneumothorax;
* Presenting a first episode of pneumothorax spontaneous primary with risk factor of recurrence
* The unsticking must be complete or important (superior to 3 cms between the summit of the lung and the summit of the thoracic cavity or superior to 2 cms with regard to the side thoracic wall);
* Benefiting from a national insurance scheme;
* Agreeing to participate in the study, and having read, included and signed the note of information intended in patients.

Exclusion Criteria:

* Subjects:Presenting a traumatic pneumothorax; Presenting a pneumothorax iatrogÃƒÂ¨ne; Presenting a secondary spontaneous pneumothorax ( underlying pleuro-lung pathology); Presenting bubbles of emphysema of size(cutting) superior to 5 cms; presenting a pneumothorax catamenial;Presenting one of the following concomitant severe pathologies dissuading a general anesthetic or any symphysant gesture(movement): cardiac insufficiency
* Pregnant or breast-feeding Woman;
* presenting neurological disorders or psychiatric forbidding the understanding of the essay;
* Who the follow-up is impossible;
* Deprived of freedom following a court or administrative order;
* Not having signed the enlightened assent.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2009-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
to show the non-inferiority of talc pleurodesis under medical thoracoscopy versus pleurodesis under video-assisted thoracoscopy surgery for recurrent primary spontaneous pneumothorax | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne FRATICELLI, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Service d'Oncologie Thoracique- HÃ´pital Sainte Marguerite, Marseille, France